CLINICAL TRIAL: NCT03684460
Title: Daytime Bright Light, Circadian Abnormalities, and Delirium in Medical ICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000023033; 000 (Other: CTGTY)
Record Dates: First submitted 2018-06-05; First posted 2018-09-25 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Circadian Rhythm Disorders
Keywords: circadian misalignment; bright light; entrainment; zeitgeber; critical illness; delirium; actigraphy
MeSH Terms: conditions — Chronobiology Disorders; Critical Illness; Delirium

STUDY DESIGN:
Intervention Model Description: randomized controlled trial with 2 cohorts
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bright Light (Experimental): Intervention: Daytime Bright Light
  Patients will be eligible if they were admitted within 30 hours of noon on enrollment day (e.g. at or after 06:00 on the prior calendar day). Enrollment will occur before noon, and the day of enrollment is termed study day 1.
  Patients will undergo monitoring (light levels, circadian alignment), starting on study day 1. Patients will be exposed to bright light from 09:00 to 13:00 starting on study day 2 and continuing through study day 5 or MICU discharge whichever is longer up to 30 days. Bright light exposure will occur in the Intensive Care Unit (ICU) and on the floor, if the patient is transferred (prior to study day 5). Feasibility metrics will also be collected.
  Interventions: Device: Daytime Bright Light
- Usual Light (Active Comparator): Intervention: Usual Care
  Patients will be eligible if they were admitted within 30 hours of noon on enrollment day (e.g. at or after 06:00 on the prior calendar day). Enrollment will occur before noon, and the day of enrollment is termed study day 1.
  Patients will undergo monitoring (light levels, circadian alignment), but otherwise, have usual care.
  Interventions: Device: Usual Light

INTERVENTIONS:
Device: Daytime Bright Light — Daytime Bright Light (DBL) will be delivered by a free-standing apparatus set to deliver 10,000 lux. The device will be placed at the bedside within 36 inches of the patient's head and is expected to provide at least 1,250 lux at the angle of gaze. To remain in the study, the patient must be in the Intensive Care Unit (ICU) through 13:00 on day 2 (e.g., the first day of potential intervention). After day 2, DBL and other study activities will continue if the patient is transferred out of the ICU to the general medical floor.
  Arms: Bright Light
Device: Usual Light — Usual care lighting in ICU.
  To remain in the study usual care patients must also remain in the MICU through 13:00 on day 2.
  Arms: Usual Light

SUMMARY:
To determine if daytime bright light will promote circadian alignment and shorten or prevent delirium.

DETAILED DESCRIPTION:
To determine if daytime bright light will promote circadian alignment and shorten or prevent delirium. The objective is to conduct a randomized controlled trial to determine if a circadian entrainment intervention, daytime bright light, will promote circadian alignment and reduce days of delirium

ELIGIBILITY:
Inclusion Criteria:

1. Hospital admission ≤30 hours at noon on enrollment day
2. Expected to say in the Medical Intensive Care Unit (MICU) ≥24 hours after enrollment
3. Age ≥50 years

Exclusion Criteria:

1. At significant risk for pre-existing circadian abnormalities:

   * Severe chronic brain injury (Injury greater than 30 days ago resulting in the inability to live independently)
   * Acute brain injury of any severity (Injury less than 30 days ago including acute intracranial bleed, traumatic brain injury, central nervous system infection, tumor)
   * Documented circadian disorder or blind/disease of the optic nerve
   * Current history of substance abuse including alcohol (use in last 30 days)

3. Transferred from an outside hospital. 4. History of bipolar disease 5. Paralyzed (due to injury, disease or medications)

Enrolled patients who do not stay in the MICU through 13:00 of Study Day 2 will be excluded; patients transferred from the MICU to the floor between 22:00 and 05:00 on subsequent study nights will continue in the study but be excluded from the primary analysis (estimated 10% of patients).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Circadian Alignment | Study Day 1-30 (to study day 5 or MICU discharge whichever is longer, patients will be censored at hospital discharge).
  The primary circadian outcome will be the proportion of daytime activity out of total activity (daytime proportion). Rest-activity patterns will be measured with the Actiwatch Spectrum (Philips Healthcare, Netherlands) set at 30-second epochs and placed on the patient's wrist.
  Enrolled patients who do not stay in the MICU through 13:00 of Study Day 2 will be excluded from all analysis.
Days of Delirium | Study Day 1-30 (patients will be censored at hospital discharge)
  The approach is to measure days of delirium in our patient cohort. After enrollment, the investigators will check patients daily for delirium until hospital discharge or day 30.

SECONDARY OUTCOMES:
Circadian Alignment, Secondary Measures, Body surface temperature gradient | Study Day 1-30 (to study day 5 or MICU discharge whichever is longer, patients will be censored at hospital discharge).
  The investigators will include additional measures of circadian alignment in our analysis: continuous body surface temperature gradient.
Circadian Alignment, Secondary Measures, Continous Heart Rate | Study Day 1-30 (to study day 5 or MICU discharge whichever is longer, patients will be censored at hospital discharge).
  The investigators will include additional measures of circadian alignment in our analysis: continuous heart rate.
Circadian Alignment, Secondary Measures, urinary 6-sulfatoxymelatonin. | Study Day 1-30 (to study day 5 or MICU discharge whichever is longer, patients will be censored at hospital discharge).
  The investigators will include additional measures of circadian alignment in our analysis: urinary 6-sulfatoxymelatonin (for patients making sufficient urine and with an indwelling urinary catheter).
Feasibility, Patient Acceptance | Study Day 1
  Percent of patients/surrogates who agree to bright light when initially described to them.
Feasibility, Patient Tolerance Time | Study Day 2-30 (to study day 5 or MICU discharge whichever is longer, patients will be censored at hospital discharge).
  Percent of intended treatment hours that patient continues with the delivery of bright light once exposed to bright light.
Feasibility, Patient Tolerance Symptoms | Study Day 2-30 (to study day 5 or MICU discharge whichever is longer, patients will be censored at hospital discharge).
  Percent of patients who develop eyestrain, headache or visual disturbance (combined outcome).
Feasibility, Intervention Fidelity | Study Day 2-30 (to study day 5 or MICU discharge whichever is longer, patients will be censored at hospital discharge).
  Percent of time per day that device delivers the planned dose of light.
Feasibility, Intervention Sustainability | Study Day 2-30 (to study day 5 or MICU discharge whichever is longer, patients will be censored at hospital discharge).
  Percent of intended intervention days that the device is used. For this metric, days that the patient refuses bright light will not be included in "intended intervention days."
Total Sleep | Study Day 1-30 (to study day 5 or MICU discharge whichever is longer, patients will be censored at hospital discharge).
  The investigators will measure (and control for) the total amount of sleep (sleep quantity) via actigraphy.
Sleep Efficiency | Study Day 1-30 (to study day 5 or MICU discharge whichever is longer, patients will be censored at hospital discharge).
  The investigators will measure (and control for) overnight sleep efficiency (sleep quality) via actigraphy.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Knauert, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, York Street Campus, New Haven, Connecticut, United States